CLINICAL TRIAL: NCT02747368
Title: Evaluation of Visual Function and Driving Health Using Ocusweep in Patients Suffering From Wet Age-related Macular Degeneration
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Turku University Hospital (Other Government)
Responsible Party: Principal Investigator, Vesa Aaltonen, Consultant in Ophthalmology, Turku University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: T220/2015
Record Dates: First submitted 2016-04-08; First posted 2016-04-21 (Estimated); Last update posted 2017-04-26 (Actual); Status verified 2017-04

CONDITIONS: Macular Degeneration
Keywords: Wet age-related macular degeneration; Age-related macular degeneration; Ocusweep; Driving health; Visual field; Contrast sensitivity
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Wet age related macular degeneration (Other): Ocusweep system is compared to results of conventional devices.
  Interventions: Device: Ocusweep system

INTERVENTIONS:
Device: Ocusweep system — Comparison of Ocusweep system to conventional visual acuity, contrast sensitivity and visual field testing.

SUMMARY:
The aim is to study the use of Ocusweep system especially in driving health evaluation and compare the results produced by Ocusweep system to those of conventional devices. The main focus is in patients suffering from wet age-related macular degeneration. The study aims to find out how frequently these patients do not meet the European Union health criteria of safe driving and how Ocusweep finds these patients from a population of patients being treated in a busy medical retina clinic. The tests of Ocusweep system are compared against conventional visual field tests, contrast sensitivity tests, visual acuity tests and tests showing anatomical changes related to wet age-related macular degeneration (optical coherence tomography, fundus photography and fluorescein or indocyanine green angiography).

ELIGIBILITY:
Inclusion Criteria:

* Macular degeneration or other diagnosed or suspected macular disease

Exclusion Criteria:

* Pregnancy
* Mental disorder
* Dementia and Alzheimers disease
* Prisoners

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2016-04; Primary Completion 2021-04 (Estimated); Study Completion 2021-04 (Estimated)

PRIMARY OUTCOMES:
Evidence that Ocusweep finds patients not meeting health criteria for driving, measured by absolute scotoma in central visual field | 2 years
Evidence that Ocusweep finds patients not meeting health criteria for driving, measured by narrowing of peripheral visual field | 2 years
Evidence that Ocusweep finds patients not meeting health criteria for driving, measured by visual acuity score | 2 years
Evidence that Ocusweep finds patients not meeting health criteria for driving, measured by contrast sensitivity score | 2 years
Evidence of whether Ocusweep is comparable to conventional methods or not, by comparison of results acquired by central visual field testing | 4 years
Evidence of whether Ocusweep is comparable to conventional methods or not, by comparison of results acquired by peripheral visual field testing | 4 years
Evidence of whether Ocusweep is comparable to conventional methods or not, by comparison of results in visual acuity scores | 4 years
Evidence of whether Ocusweep is comparable to conventional methods or not, by comparison of results in contrast sensitivity score | 4 years
Evidence which (Ocusweep or ophthalmologist) is better in finding patients not meeting health criteria for driving, by comparison of results acquired by central visual field testing | 2 years
Evidence which (Ocusweep or ophthalmologist) is better in finding patients not meeting health criteria for driving, by comparison of results acquired by peripheral visual field testing | 2 years
Evidence which (Ocusweep or ophthalmologist) is better in finding patients not meeting health criteria for driving, by comparison of results in visual acuity scores | 2 years
Evidence which (Ocusweep or ophthalmologist) is better in finding patients not meeting health criteria for driving, by comparison of results in contrast sensitivity score | 2 years

IPD SHARING:
Plan to Share IPD: No